CLINICAL TRIAL: NCT01532609
Title: Methadone Maintenance and HIV Prevention: A Window of Opportunity in China Version
Brief Title: Methadone Maintenance and HIV Prevention: A Window of Opportunity in China
Acronym: MMT1
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Los Angeles (Other)
Collaborators: Centers for Disease Control and Prevention, China (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: R34MH083512 (NIH)
Record Dates: First submitted 2012-02-08; First posted 2012-02-14 (Estimated); Last update posted 2023-10-02 (Actual); Status verified 2023-09

CONDITIONS: Capacity Building; Drug Use; HIV/AIDS
Keywords: Methadone maintenance therapy; Behavioral intervention; Service provider; Drug use
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Intervention (Experimental): Intervention group service providers received four training sessions (plus reunion sessions) on MMT protocol, reducing stigma and its impact, maintaining positive interactions with clients, and motivational interviewing skills. The participating providers are required to conduct three individual motivational sessions with their clients upon completion of the intervention sessions.
  Interventions: Behavioral: MMT CARE
- Standard care (No Intervention): No additional training or service is provided for standard care group service providers or clients.

INTERVENTIONS:
Behavioral: MMT CARE — Intervention group service providers received four training sessions (plus reunion sessions) on MMT protocol, reducing stigma and its impact, maintaining positive interactions with clients, and motivational interviewing skills. The participating providers are required to conduct three individual motivational sessions with their clients upon completion of the intervention sessions.
  Arms: Intervention

SUMMARY:
This study is an intervention pilot that integrates the current methadone maintenance treatment (MMT) program in China with psychosocial and behavioral components in order to address the critical link between drug use and HIV/AIDS.

The intervention pilot proceeds in two phases in Sichuan, China. In Phase 1, we developed the intervention manuals and supporting materials, and finalized assessment measures and implementation procedures. In Phase 2, we conducted an intervention pilot across 6 MMT clinics involving 41 service providers and 179 clients, and followed up at three, six, and nine months.

DETAILED DESCRIPTION:
The implementation of the MMT program in China is one of the most significant measures ever taken by the Chinese government to address drug use and HIV prevention challenges. In 2004, China launched a series of MMT programs at eight pilot clinics in five provinces. By December 2007, 503 MMT clinics had been established nationwide across 23 provinces. Several studies have found that positive outcomes in drug use, criminality, and employment were associated with participation in MMT. However, special challenges are facing the current MMT programs are facing: 1) clients' drop-out rates are high; and 2) providers at MMT clinics do not have sufficient training, and some of them hesitate to serve the population. We have recognized the urgent need and conducted the study to address these challenges.

The intervention pilot proceeds in two phases in Sichuan, China. In Phase 1, we developed the intervention manuals and supporting materials, and finalized assessment measures and implementation procedures. In Phase 2, we conducted an intervention pilot across 6 MMT clinics involving 41 service providers and 179 clients, and followed up at three, six, and nine months.

The specific aims of the proposed study are:

Specific Aim 1: To assess the feasibility and acceptability of the MMT PLUS intervention with process evaluation and participant feedback.

Specific Aim 2: To examine primary outcomes on whether service providers in the intervention group, compared to providers in the standard care, will demonstrate improved adherence to MMT protocol, decrease in prejudicial attitudes, increase in comfort working with MMT clients, increase in motivating clients and making personalized risk management plan.

Specific Aim 3: To explore secondary outcomes on whether MMT clients in the intervention group, compared to clients in the standard care, will report increased motivation to change, improved psychological and physical health, increased positive support network, and reduced HIV risk behavior.

Specific Aim 4: To investigate exploratory outcomes on whether MMT clients in the intervention group, compared to clients in the standard care, will report improved MMT treatment retention and decreased drug use.

ELIGIBILITY:
Inclusion Criteria:

Service providers

* Age 18 and above
* Currently working in MMT clinic
* Informed consent

MMT clients

* Age 18 or over
* Currently enrolled in MMT
* Informed consent

Exclusion Criteria:

Service providers

* Anyone who does not meet the inclusion criteria.

MMT clients:

* Psychosis, neurological damage, as judged by an interviewer in consultation with a clinical supervisor inability to give informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 220 (Actual)
Dates: Start 2009-03; Primary Completion 2010-12 (Actual); Study Completion 2011-03 (Actual)

PRIMARY OUTCOMES:
Service providers' MMT knowledge | Changes from baseline to 3-, 6- and 9-month follow-up
Service provider's prejudical attitude towards drug users | Changes from baseline to 3-, 6- and 9-month follow-up
Provide-client interaction | Changes from baseline to 3-, 6- and 9-month follow-up
Provider's perceived stigma due to work with drug using population | Changes from baseline to 3-, 6- and 9-month follow-up
Service provider's perceived risk at work | Changes from baseline to 3-, 6- and 9-month follow-up
Service provider's perceived institutional support | Changes from baseline to 3-, 6- and 9-month follow-up
Service provider's job satisfaction | Changes from baseline to 3-, 6- and 9-month follow-up

SECONDARY OUTCOMES:
Client's drug using behavior | Changes from baseline to 3-, 6- and 9-month follow-up
Client's physical health | Changes from baseline to 3-, 6- and 9-month follow-up
MMT client's mental health | Changes from baseline to 3-, 6- and 9-month follow-up
Client's perceived stigma from MMT clients | Changes from baseline to 3-, 6- and 9-month follow-up
Client's readiness to change | Changes from baseline to 3-, 6- and 9-month follow-up
Client's drug avoidance self-efficacy | Changes from baseline to 3-, 6- and 9-month follow-up
Client's social support | Changes from baseline to 3-, 6- and 9-month follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Li Li, PhD, Principal Investigator — NPI-Center for Community Health, UCLA
Locations (1):
- Sichuan Provincial Center for Disease Control and Prevention, Chengdu, Sichuan, China

REFERENCES:
- [Derived] Li L, Wu Z, Liang LJ, Lin C, Zhang L, Guo S, Rou K, Li J. An intervention targeting service providers and clients for methadone maintenance treatment in China: a cluster-randomized trial. Addiction. 2013 Feb;108(2):356-66. doi: 10.1111/j.1360-0443.2012.04020.x. Epub 2012 Oct 5. PMID 22788780